CLINICAL TRIAL: NCT01596803
Title: Effects of Antioxidants Supplementation on Muscular Function of Patients Affected by Facioscapulohumeral Dystrophy (FSHD)
Brief Title: Effects Antioxidants Supplementation on Muscular Function Patients Facioscapulohumeral Dystrophy (FSHD)
Acronym: FSHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Hospital Clinical Research Project 2010 (Unknown); Association Amis FSH France (Unknown); FSH Dutch Fondation The Netherland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 8426
Record Dates: First submitted 2012-04-05; First posted 2012-05-11 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
Keywords: FSHD; Antioxidants; Oxidative stress; Muscle function; Quality of life; Activity; (FSHD;4q35)
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Motor Activity | interventions — Antioxidants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamins minerals (Active Comparator): VitE 400/d, vitC 500mg/d, Se 200µg/d (selenomethionine), Zn 25 mg/d gluconate Venous blood samples( analysis oxidative stress inflammatory markers) Needle biopsy of the vastus lateralis muscle (analysis oxidative stress inflammatory markers)
  Interventions: Procedure: Taking of blood; Dietary Supplement: needle biopsy of the vastus lateralis muscle; Dietary Supplement: Vit C Vit E Zn Se
- Placebo (Placebo Comparator): Supplementation 17 weeks placebo venous blood samples (analysis of oxidative stress inflammatory markers) needle biopsy of the vastus lateralis muscle
  Interventions: Procedure: Taking of blood; Dietary Supplement: needle biopsy of the vastus lateralis muscle; Dietary Supplement: Placebo Vit E Placebo Vit C Zn Se

INTERVENTIONS:
Procedure: Taking of blood — Taking venous blood samples to analyse oxidant stress
Dietary Supplement: needle biopsy of the vastus lateralis muscle — T0 needle biopsy of the vastus lateralis muscle (analysis of oxidative stress and inflammatory markers)During 17 weeks supplementation by Vit E, C , Zn Se After 17 weeks: veinous blood samples and needle biopsy
Dietary Supplement: Vit C Vit E Zn Se — T0 venous blood samples and needle biopsy of the vastus lateralis muscle During 17 weeks vit E 400mg/d, Se 200µg/d, Vit C 500mg/day, Zn 25 mg/d After the supplementation of 17 weeks:venous blood samples and needle biopsy of the vastus lateralis muscle
  Other Names: FSHD; Antioxidant
  Arms: vitamins minerals
Dietary Supplement: Placebo Vit E Placebo Vit C Zn Se — venous blood samples and needle biopsy
  Arms: Placebo

SUMMARY:
On the basis of published data and the investigators' results indicating that oxidative stress may contribute to the peripheral skeletal muscle dysfunction in patients with FSHD, the investigators propose a study to test whether or not an antioxidant supplementation has a therapeutic interest for patients with FSHD. Their results have important implications for the successful implementation of rational antioxidant therapy in FSHD in which cell loss could be linked to oxidative stress.

DETAILED DESCRIPTION:
This study will compare the effect of the therapeutic interest of an antioxidant supplementation on the functional deficits and the molecular muscle abnormalities into two groups of patients affected by FSHD, one treated with the antioxidant supplementation during 17 weeks. The antioxidant by capsule consisted of:Vitamin E (400 mg /day), Selenium (200 µg/day in the form of selenomethionine), Vitamin C (500 mg/day), Zinc (25 mg/day in the form of gluconate). The second one treated with a placebo during 17 weeks. Patients will be assigned to intervention groups by chance, and neither physician, nor patient, will know which product is administrated (study in "double blind").

ELIGIBILITY:
Inclusion Criteria:

* FSHD patients will be recruited on the basis of:

  * The number of repeat units (4 to 9)
  * FSHD patients with a positive family history for FSHD
  * Not confined to a wheelchair
  * No smokers
  * No associated co-morbidity (cardiac or pulmonary disease, diabetes etc.)
  * No Medications or nutritional supplementation (vitamins and/or antioxidants) at the time of the study
  * No HIV positive

Exclusion Criteria:

* No consent form

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2012-02-20 (Actual); Study Completion 2012-06-01 (Actual)

PRIMARY OUTCOMES:
Improvement of muscle effort tolerance after antioxidant supplementation | duration study 3 years
  17-weeks evaluation of an antioxidant supplementation in order to modulate or delay oxidative insult that could be useful to maintain FSHD muscle function. At T0, each patient will perform functionnal evaluation (Exercise Tolerance (2 minutes walking test), and/or Maximal Volontary Contraction and/or Endurance of quadriceps muscles).

SECONDARY OUTCOMES:
Changes in inflammatory and oxidative stress parameters after antioxidant supplementation | duration study 3 years
  T0 evaluations spirometry, electrocardiogram, holter,Magnetic Resonance imaging of the both thighs,estimation muscle oxygen consumption during acute exercise . T7 venous blood samples (oxidative stress inflammatory markers)needle biopsy of the vastus lateralis muscle (oxidative stress inflammatory markers). analysis oxidative stress on muscle biochemical analyses.T7 patient receives placebo or antioxidant supplementation corresponding randomly-assigned trial. After 17 weeks supplementation the subjects will obtain venous blood samples and needle biopsy.
Changes in muscular function after antioxidant supplementation | duration study 3 years
  T0 evaluations spirometry, electrocardiogram, holter Magnetic Resonance imaging of the both thighs,estimation muscle oxygen consumption . T7 venous blood samples (oxidative stress inflammatory markers)needle biopsy of the vastus lateralis muscle (oxidative stress inflammatory markers). This one-week lap's time is needed to avoid potential confounding effects of exercise-induced oxidative stress on muscle biochemical analyses.T7 patient receives placebo or antioxidant supplementation corresponding randomly-assigned trial. After 17 weeks supplementation venous blood samples and needle biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital- Saint Eloi Hospital, Montpellier, Languedoc-Roussillon, France

REFERENCES:
- [Derived] Passerieux E, Hayot M, Jaussent A, Carnac G, Gouzi F, Pillard F, Picot MC, Bocker K, Hugon G, Pincemail J, Defraigne JO, Verrips T, Mercier J, Laoudj-Chenivesse D. Effects of vitamin C, vitamin E, zinc gluconate, and selenomethionine supplementation on muscle function and oxidative stress biomarkers in patients with facioscapulohumeral dystrophy: a double-blind randomized controlled clinical trial. Free Radic Biol Med. 2015 Apr;81:158-69. doi: 10.1016/j.freeradbiomed.2014.09.014. Epub 2014 Sep 20. PMID 25246239